CLINICAL TRIAL: NCT03426137
Title: Relieving Acute Pain (RAP): A Pilot Study
Brief Title: Relieving Acute Pain (RAP) Study: A Pilot Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The focus of the project has shifted to publishing a protocol for future trials because we were unable to recruit. Three participants signed the consent forms but withdrew before the randomization.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Luana Colloca, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00078742
Record Dates: First submitted 2018-01-16; First posted 2018-02-08 (Actual); Results first posted 2020-03-16 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Trauma; Opioid Use; Spine Fusion
Keywords: Oxycodone; Placebo; Expectancy Induced Analgesia; NSAID
MeSH Terms: conditions — Wounds and Injuries | interventions — Oxycodone; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to three arms. Arm 1 will be a Full Dose (FD) group, which will receive all NSAIDs will be dosed in accordance with the STC Guidelines for NSAID use and Oxycodone (5mg). Arm 2 will be a Partial Reinforcement (PR) group, which will receive NSAIDs, Oxycodone (5mg), and placebo pills to reach a 50% reduction of the total intake of opioids. Finally, Arm 3 will be a Control (C) group receiving NSAIDs and placebos.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Oxycodone and Placebo will be identical in terms of appearance, taste, and smell so as to keep the investigators, care providers, and participants blind to their treatment allocation. Oxycodone and placebo oral suspensions will be manufactured and dispensed by the pharmacy at University of Maryland Medical Center. All research personnel, aside from the pharmacists and team members responsible for final review and write-up of the study, will be blinded to participants' treatment groups. For participants in the Partial Reduction group (Arm 2), the pharmacy will dispense the study drug such that participants in Arm 2 will receive four doses of Oxycodone (5mg) followed by one of four repeating schedules of administration alternating between Oxycodone (5mg) and placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Full Dose (FD) (Active Comparator): Participants in the FD arm will receive NSAIDs and Oxycodone (5mg).dosed in accordance with the Guidelines for Use from University of Maryland Shock Trauma Center.
  Interventions: Drug: Oxycodone; Drug: Ketorolac
- PR (Partial Reinforcement) (Placebo Comparator): Participants in this group will receive NSAIDs, Oxycodone (5mg), and placebo pills to reach a 50% reduction of the total intake of opioids.
  Interventions: Drug: Oxycodone; Drug: Ketorolac; Other: Placebo
- C (Control) (Placebo Comparator): Participants in this group will receive NSAIDs and placebo pills
  Interventions: Drug: Ketorolac; Other: Placebo

INTERVENTIONS:
Drug: Oxycodone — 5mg Oxycodone in oral solution given every 3 hours
  Other Names: Oxycodone Hydrochloride
  Arms: Full Dose (FD); PR (Partial Reinforcement)
Drug: Ketorolac — toradol intravenous (IV) 30mg. Maintain toradol IV every 8 hours, round the clock. For patients with renal insufficiency, decrease toradol dose to 15mg every 8 hours. For patients over 65 years old, decrease toradol dose to 15 mg every 8 hours. After 24 hours, start oral NSAIDS every 8 hours round the clock when tolerating pain.
  Other Names: Toradol
Other: Placebo — Oral solutions containing only the carrier vehicle - a flavored syrup called OraSweet
  Other Names: OraSweet
  Arms: C (Control); PR (Partial Reinforcement)

SUMMARY:
The United States (US) faces a crisis of pain management. According to the 2012 National Health Interview Survey, almost 50 million adults in the US reported having significant chronic or severe pain (Nahin 2015). Doctors in the US still prescribe opioids across the board for pain despite a growing recognition of an epidemic of opioid overdose and use disorder. Few solutions have been successfully proposed and implemented. Placebos represent a novel and potentially fruitful means of addressing this issue. However, clinicians often use placebos deceptively and with little rationale or evidence of benefit, making their use ethically problematic. In contrast with their typical current use, a provocative line of research suggests that placebos can be intentionally exploited to extend analgesic therapeutic effects. Recently, we reviewed a database of placebo studies including 22 studies in both animals and humans hinting of evidence that placebos may work as a dose extender of active painkillers. Placebos given after repeated administration of active treatments can acquire medication-like effects based on learning mechanisms.

Here, we will test if dose-extending placebos are effective in relieving clinical acute pain in opioid patients with traumatic pain. Patients will be randomized to three arms. Arm 1 will be a Full Dose (FD) group, which will receive all NSAIDs as described in the Guidelines for NSAID use in Orthopedic Patients and Oxycodone (5mg). Arm 2 will be a Partial Reinforcement (PR) group, which will receive NSAIDs, Oxycodone (5mg), and placebos to reach a 50% reduction of the total intake of opioids. Finally, Arm 3 will be a Control (C) group receiving NSAIDs and placebos. Patients will be assigned to one of three arms according to a 1:1:1 schedule of randomization. Study IDs will be generated by the pharmacy and blinding will occur by ensuring that oxycodone and placebos look, smell, and taste identical. Rescue therapy will be provided as needed. This novel prospect of placebo use has the potential to change our general thinking about painkiller treatments, the typical regimens of painkiller applications, and the ways in which treatments are evaluated.

DETAILED DESCRIPTION:
Overview:

We will screen 500 patients from the Shock Trauma Center to recruit a total of 159 (53 per arm) to participate in a pilot study aimed at reducing use of opioids. Participants will meet all of the eligibility criteria and none of the exclusion criteria. After enrollment, participants will be blindly allocated to one of three randomization arms by means of de-identified Study IDs corresponding to treatment arms. Study IDs will be generated by the pharmacy and blinding will be ensured by creating study drugs that look, smell, and taste identical. The pharmacy will create and dispense identical study drugs in terms of appearance, smell, and taste. Only the blinding coordinator will know the identity of patients in each treatment arm. Arm 1 will be a Full Dose (FD) group, which will receive Non-Steroidal Anti-Inflammatory Drugs (NSAIDs), dosed in accordance with the University of Maryland Shock Trauma Center (STC) Guidelines for NSAIDs and Oxycodone (5mg). Arm 2 will be a Partial Reinforcement (PR) group, which will receive NSAIDs, Oxycodone (5mg), and placebos to reach a 50% reduction of the total intake of opioids. Finally, Arm 3 will be a Control (C) group receiving NSAIDs and placebos. Patients will be assigned to one of these three arms according to a 1:1:1 schedule of randomization. The patient will start receiving study medication as part of his or her pain management as soon as possible after admission to the hospital and enrollment in the study (ideally as their first dose of pain-management medication). Rescue therapy will be provided as needed.

All enrolled patients will receive an Adult Pain Management Service (APMS) consult. APMS will work with the study and clinical teams to ensure that all treatment protocols are met, and be available to address any issues that may arise. The APMS provider will work with the primary service to determine the most effective NSAID as described in their guidelines.

Other than the study medication (Oxycodone and placebo), all participants will be treated in accordance with the current standard of care at the University of Maryland Shock Trauma Center. This includes intravenous Toradol every 8 hours for 24 hours followed by oral NSAIDs round the clock until pain is minimal. The timing of administration will be the same for participants in all three arms - they will receive their arm's treatment (Oxycodone, Oxycodone alternating with placebo, or no additional medication beyond standard of care NSAIDs) round the clock for the first 24 hours followed by every hours for the remainder of hospitalization. All patients will receive intravenous Dilaudid every hour for rescue or break through pain. In addition, all patients will be discharged on Oxycodone tablets (5mg) every 3 hours as needed.

In Arm 2, the first four doses of study drug will be Oxycodone (5mg) to condition them to its effects. Afterwards, they will receive alternating Oxycodone (5mg) and placebo according to one of four repeating sequences. During data analysis, we will test whether the sequence of administration has an effect on outcomes. Participants in Arm 2 will never receive more than 2 doses of placebo in a row. This administration schedule will be repeated for the remainder of hospitalization.

Prior to patients' enrollment:

The intent of this study is to enroll 159 patients with trauma into this study to compare strategies to reduce opioid use during the management of acute pain. Patients will be screened on admission to the Shock Trauma Center. Eligible patients will meet all of the inclusion criteria and none of the exclusion criteria. Patients with trauma will be considered for enrollment and be flagged for screening. A plan by the primary service to adhere to The Shock Trauma Protocol for NSAID use is also a requirement for enrollment. Eligible participants will be informed and have the opportunity to discuss the nature of the study, potential for treatment allocation, and risk/benefits. For those who agree to participate, the approved Informed Consent Form and HIPAA authorization form will be signed. The research staff will explain to the participant what tasks they are expected to complete during this study, answer any questions they may have, and ensure comprehension by completing the Informed Consent Checklist, which asks participants to verbally report their understanding of the study purpose and procedures, among other key points.

Allocation to treatment group:

After the participant discusses and signs the consent form, a staff member will call the pharmacy to inform them of the participant's de-identified Screening number. The pharmacy will then randomly assign that participant a Study ID corresponding randomly to one of the three treatment groups and handle drug logistics (sourcing, processing, and administration) for the remainder of Phase I. The patient will start receiving the study drug within 24 hours of being able to take narcotics, ideally as his/her first narcotic medication. All staff involved with the protocol will be fully trained on it and will be given study team member emergency contacts in case of incident.

Blinding:

Oxycodone and Placebo will be identical in terms of appearance, taste, and smell so as to keep both the investigators and participants blind to their treatment allocation. Oxycodone and placebo oral suspensions will be manufactured by the IDS. Oxycodone solution will be made from tablets to ensure blinding. In this way, both Oxycodone and placebo will look identical for taste, color, and smell. This will help not only to blind the study, but also facilitate study drug administration given that patients may be intubated. All research personnel, aside from the pharmacists and team members responsible for final review and write-up of the study, will be blinded to participants' treatment groups. The pharmacy will dispense medications for each participant that will correspond with their allocated treatment group. For participants in the Partial Reduction group (Arm 2), the pharmacy will dispense the study drug. In summary, participants in Arm 2 will receive four doses of Oxycodone (5mg) followed by one of four repeating schedules of administration alternating between Oxycodone (5mg) and placebo.

Hospitalization window (Enrollment - End of Hospitalization):

Pain ratings will be recorded as usual within 20 to 90 minutes after each study drug administration. Also, participants will be given the option to complete a set of psychological questionnaires during the time in the hospital or by the time of their first follow-up visit. Questionnaires unrelated to pain will be optional. Although we cannot change the wording of our validated pain questionnaires, staff will be trained to use the phrasing such as "how well they are able to perform their daily activities, how well they are able to interact with visitors/family, and how well they are sleeping" whenever possible, and that surveys andquestions during the follow-up phase will also take this non-pain-centric approach.

Discharge:

Participants will be monitored for subsequent use of opioids at the first post-discharge visit (at approximately 2 weeks) and within month 1, 3, and 6 for follow-ups. The research team via calls, letters, emails, or texts. REDCap, Qualtrics / MetricWire will be used to facilitate the communication via text and emails. The team member will ask the participant questions about their health and medication use. In addition, a phone application may be developed or the data collection system Qualtrics used to gather information about participants' medication use and health during the follow-up period. Although the wording of the validated Pain Questionnaires we will use during hospitalization cannot be changed, during the follow-up phase we will aim to frame questions about pain intensity and interference with function in such a way as to avoid nocebo effects (i.e. asking how well they are able to perform their daily activities, how well they are able to interact with visitors/family, and how well they are sleeping instead of how much pain are they experiencing).

Duration of the clinical trial:

Hospitalization window (starting as soon after admission as possible for a projected minimum of 2 days), with follow-up at approximately 2 weeks (coinciding with their first post-discharge visit with their clinician), and months 1, 3, and 6.

Rescue plan:

All patients will have the same rescue medicine available for break through pain; intravenous Dilaudid every hour.

Participants in each of the three randomization arms will have access to opioid rescue medication (Dilaudid) as needed via a standing order for breakthrough pain rated as Severe. The rate of use pf rescue therapy will be evaluated as a primary endpoints. Participants who request more than 3 doses of rescue medication in a row will be withdrawn from the study and referred to APMS for further pain management.

Primary and secondary outcomes. To be measured daily during hospitalization

1.) Acute clinical and functional pain / acute pain improvement; opioid intake; rate of request of rescue therapies.

Primary and secondary outcomes. To be measured daily during the follow-up.

1. Use (frequency and intensity) of opioid prescriptions
2. Development of dependence and/or addiction problems

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Admission to The Shock Trauma Center within 72 hrs
* Any trauma requiring inpatient opioid medication
* Plan by primary service to follow the Shock Trauma Guidelines for Acute Pain in Orthopedic Injury
* Predicted length of stay greater than or equal to 2 days

Exclusion Criteria:

* Non English speaking
* Spine cord injury
* Severe Traumatic brain injury (based on a Glascow Coma Scale of 8 or less)
* Patient-controlled analgesia
* Admission Creatinine > 1.4
* History of chronic kidney disease
* Heroin use in the 3 months prior to admission (patient self-report)
* Severe psychiatric condition (e.g. schizophrenia, bipolar disorders, mania, autism) and /or psychiatric condition leading to treatment and/or hospitalization within the last 1 year.
* Positive toxicology screen for methadone not prescribed during current hospitalization
* Pregnancy or breast feeding
* Contraindication to NSAIDs, including high risk of bleeding or known severe coronary artery disease
* Injuries deemed non survival.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2020-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luana Colloca, MD/PHD/MS, Principal Investigator — University of Maryland Baltimore School of Nursing
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared among study team members.

REFERENCES:
- [Background] Chen EY, Marcantonio A, Tornetta P 3rd. Correlation Between 24-Hour Predischarge Opioid Use and Amount of Opioids Prescribed at Hospital Discharge. JAMA Surg. 2018 Feb 21;153(2):e174859. doi: 10.1001/jamasurg.2017.4859. Epub 2018 Feb 21. PMID 29238810
- [Background] Hah J, Mackey SC, Schmidt P, McCue R, Humphreys K, Trafton J, Efron B, Clay D, Sharifzadeh Y, Ruchelli G, Goodman S, Huddleston J, Maloney WJ, Dirbas FM, Shrager J, Costouros JG, Curtin C, Carroll I. Effect of Perioperative Gabapentin on Postoperative Pain Resolution and Opioid Cessation in a Mixed Surgical Cohort: A Randomized Clinical Trial. JAMA Surg. 2018 Apr 1;153(4):303-311. doi: 10.1001/jamasurg.2017.4915. PMID 29238824
- [Background] Howard R, Waljee J, Brummett C, Englesbe M, Lee J. Reduction in Opioid Prescribing Through Evidence-Based Prescribing Guidelines. JAMA Surg. 2018 Mar 1;153(3):285-287. doi: 10.1001/jamasurg.2017.4436. PMID 29214318
- [Background] Zelcer S, Kolesnikov Y, Kovalyshyn I, Pasternak DA, Pasternak GW. Selective potentiation of opioid analgesia by nonsteroidal anti-inflammatory drugs. Brain Res. 2005 Apr 8;1040(1-2):151-6. doi: 10.1016/j.brainres.2005.01.070. PMID 15804436
- [Background] Vanegas H, Vazquez E, Tortorici V. NSAIDs, Opioids, Cannabinoids and the Control of Pain by the Central Nervous System. Pharmaceuticals (Basel). 2010 Apr 29;3(5):1335-1347. doi: 10.3390/ph3051335. PMID 27713305
- [Background] Colloca L, Lee SE, Luhowy MN, Haycock N, Okusogu C, Yim S, Raghuraman N, Goodfellow R, Murray RS, Casper P, Lee M, Scalea T, Fouche Y, Murthi S. Relieving acute pain (RAP) study: a proof-of-concept protocol for a randomised, double-blind, placebo-controlled trial. BMJ Open. 2019 Nov 11;9(11):e030623. doi: 10.1136/bmjopen-2019-030623. PMID 31719077
- See also: Dr. Luana Colloca is the Principle Investigator for this research study. More information about her background and other research can be found at this link. — http://www.nursing.umaryland.edu/directory/luana-colloca/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three participants were consented from University of Maryland Shock Trauma Center, per protocol, between 3/17/2019 to 3/30/2019. All three withdrew before randomization or starting any study procedures.
Period: Overall Study
Arm/Group | Full Dose (FD) | PR (Partial Reinforcement) | C (Control)
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The three participants who gave written consent to participate in the study and signed the HIPAA form withdrew before randomization or starting any study procedures. Therefore there is no data available to report.
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Dose (FD) | PR (Partial Reinforcement) | C (Control) | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Continuous [unit: years]
Sex: Female, Male
Race (NIH/OMB)
Pain report [unit: units on a scale]

OUTCOME MEASURES:

1. Primary Outcome: Pain Self-reports
Description: Collected on a visual analogue scale, with 0 being "no pain" and 100 being "maximum pain tolerable"
Time Frame: Day 1-7, Week 2, Months 1, 3 and 6
Population: All three participants gave written consent to participate in the study and signed the HIPAA form, but withdrew before starting any study procedures. These 3 withdrawals were handled per protocol. As is written in the consent, "You are free to withdraw your consent at any time." Therefore, there was no analyzable data collected.
Arm/Group | Full Dose (FD) | PR (Partial Reinforcement) | C (Control)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All three participants enrolled gave written consent to participate in the study and signed the HIPAA form, but withdrew before starting any study procedures.These 3 withdrawals were handled per protocol. Therefore, there was no time period over which adverse events were collected.
Description: All three participants enrolled gave written consent to participate in the study and signed the HIPAA form, but withdrew before starting any study procedures.These 3 withdrawals were handled per protocol. Therefore, there were no participants at risk for Serious Adverse Events, All-Cause Mortality, or any Other (Not Including Serious) Adverse Events.
Arm/Group | Full Dose (FD) | PR (Partial Reinforcement) | C (Control)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Early termination due to logistical and funding issues, which lead to no analyzable data. A protocol paper has been published should other investigators wish to use the study design (DOI: 10.1136/bmjopen-2019-030623).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT03426137/Prot_ICF_001.pdf